Effect of Patient
Priorities Care
Implementation in
Older Veterans
with Multiple
Chronic Conditions

NCT04922320

January 30, 2015



# Michael E. DeBakey VA Medical Center 2002 Holcombe Boulevard (152) Houston, TX 77030

#### Dear

Thank you for your participation in the Patient Priorities Care research study with Dr. Lilian Dindo at the Michael E. DeBakey VA Medical Center in Houston.

### **Purpose**

The study will compare the usual way primary care providers make treatment decisions for patients who have multiple chronic conditions with an approach that uses patients' health priorities to guide those treatment decisions. The study will evaluate which approach may benefit Veterans the most. We are assessing how current providers use and understand the patient priorities approach.

#### **Procedures**

Our conversation should last about 20-30 minutes. You can stop the interview at any time. The interview will take place virtually over the phone or video conference. You can skip any questions that you don't want to answer. Everything you say is confidential. There is no way to tie anything you say directly back to you. Taking part in this interview, or choosing to not take part, will have no impact on your relationship with the VA. If you agree, your answers will be recorded using a digital voice recorder and transcribed.

#### **Possible Benefits & Risks**

This research may or may not benefit you directly, however, because of taking part in this study, you may learn more about the patient priorities approach. Your participation will also indirectly benefit provider workflow and patient care as this study implements a potential improvement to both workflow and patient care. The risks of doing this study are small. Some people may find it uncomfortable answering questions about their health. There is a risk of loss of confidentiality if information about you from your participation becomes known to persons outside this study, but the researchers will do everything they can to avoid that. Study materials will not be accessed by anyone outside of the research team. Your information will be stored on a secure drive accessed only by research team members in accordance with VA privacy protocols. There will be no compensation provided for your participation in this study.

## **Privacy & Confidentiality**

To protect your privacy, we will only collect information that is needed for this research. The researchers are required to keep all study information confidential and private to the extent of the law. Examples of information that we are legally required to report include abuse of a child or elderly person, or certain reportable diseases. Your participation will in no way affect your relationship standing with VA.

#### **Voluntary Participation**

Participation in this study is completely voluntary. You may choose not to participate, to end participation at any time for any reason, or to refuse to answer any individual question at any time without penalty. If you choose not to participate or if you withdraw it will not harm your relationship with your doctor or MEDVAMC. By providing verbal consent, you have not given up any of your legal rights.

### **Funding Information**

This study has been funded by VA Health Services Research and Development.

If you have questions about the research, you can contact Tracey Rosen, the Project Coordinator, at 713-794-8601 ext. 10280 or Dr. Lilian Dindo, the Principal Investigator, at 713-440-4637. If you have any

Version Date: January 30, 2015

questions about your rights as a subject, you may contact the Institutional Review Board for Baylor College of Medicine and Affiliated Hospitals (IRB) at 713-798-6970. If you have any complaints, concerns, or pertinent questions regarding the conduct of this study, you may contact the investigator, Dr. Lilian Dindo, at 713-440-4637

Thank you very much for giving us some of your valuable time. We look forward to working with you.

Sincerely,

Lilian Dindo, PhD

Lilian Dindo

Version Date: January 30, 2015